#### NCT03858517

# **ReUnion TSA Statistical Analysis Plan (SAP)**

**CLINICAL INVESTIGATION** 

TITLE:

A Post-Market Clinical Evaluation of the ReUnion TSA

System

**DEVICE NAME:** ReUnion TSA System

STATISTICAL ANALYSIS PLAN

(SAP) VERSION:

2

CLINICAL INVESTIGATION

PLAN (CIP) VERSION:

1

**INDICATIONS:** This study will adhere to the indications and contraindications

for the ReUnion TSA System as are detailed in the device's

Instructions for Use.

**CLINICAL INVESTIGATION** 

**DESIGN:** 

Post-Market

• Multicenter

Prospective

• Non-Randomized

CONFIDENTIALITY STATEMENT:

This Statistical Analysis Plan contains confidential information and its' use is limited to investigational staff intending to

conduct the clinical investigation, Institutional Review Boards (IRBs)/Ethics Committees (ECs) and any others charged with

reviewing the clinical investigation.

**DATE:** 28 May 2021

# **Approval Page**

| APPROVERS | | | |
|---|---|---|---|
| Role | Name | Signature | Date |
| Author | Sascha Lorenzen | Electronically sign<br>by: Sascha<br>Lorenzen<br>Reason: I am<br>signing as the<br>Author of this<br>document<br>Sascha Lorenzen Date: May 28, 202<br>13:50 GMT+2 | 28-May-2021 |
| Statistician | Claudia Beimel | Electronically<br>signed by: Claud<br>Beimel<br>Reason: I appro-<br>this document<br>Date: May 28,<br>Claudia Beimel 2021 14:37<br>GMT+2 | |
| Clinical Research<br>Head (CRH) | Rebecca Gibson | Electronically signed by: Rebecca Gibsor Reason: I approve this document Rebecca Gibson Date: May 28, 2021 08:31 EDT | 28-May-2021 |
| Clinical<br>Investigation<br>Manager (CIM) | Susanne Höfer | Electronically<br>signed by:<br>Susanne Höfer<br>Reason: I appro<br>this document<br>Date: May 28,<br>2021 15:30<br>Susanne Höfer GMT+2 | <sup>ve</sup> 28-May-2021 |

# **Table of Contents**

| 1. | Admini | istrative Information | 5 |
|----|---------|----------------------------------------------------|----|
| | 1.1. | LIST OF ABBREVIATIONS | 5 |
| | 1.2. | STATISTICAL ANALYSIS PLAN REVISION HISTORY | 5 |
| | 1.3. | ROLES AND RESPONSIBILITIES | 6 |
| 2. | Introdu | ıction | 6 |
| | 2.1. | BACKGROUND AND RATIONALE | 6 |
| | 2.2. | CLINICAL INVESTIGATION DESIGN | 6 |
| 3. | Researc | ch Goals | 6 |
| | 3.1. | FRAMEWORK | 6 |
| | 3.2. | SAMPLE SIZE | 8 |
| 4. | Method | ls | 11 |
| | 4.1. | RANDOMIZATION | 11 |
| | 4.2. | STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE | 11 |
| | 4.3. | TIMING OF FINAL ANALYSES | |
| | 4.4. | TIMING OF OUTCOME ASSESSMENT | 11 |
| | 4.5. | STATISTICAL SOFTWARE | 12 |
| | 4.6. | MISSING DATA | 12 |
| | 4.7. | CONFIDENCE INTERVALS AND P-VALUES | 12 |
| | 4.8. | UNITS | 13 |
| | 4.9. | CALCULATIONS AND TRANSFORMATIONS | 13 |
| | 4.10. | ASSUMTIONS | 13 |
| 5. | Populat | tion and Progress | 13 |
| | 5.1. | ANALYSIS POPULATION | 13 |
| | 5.2. | ELIGIBILITY | 14 |
| | 5.3. | WITHDRAWAL / FOLLOW-UP | 14 |
| | 5.4. | ADHERENCE AND CIP DEVIATIONS | 14 |
| 6. | Analysi | is | 15 |
| | 6.1. | HARMS AND SAFETY | 15 |
| | 6.2. | BASELINE CHARACTERISTICS | 16 |
| | 6.3. | INTRAOPERATIVE CHARACTERISTICS | 20 |
| | 6.4. | EARLY POSTOPERATIVE CHARACTERISTICS | 21 |
| | 6.5. | POSTOPERATIVE CHARACTERISTICS | 22 |
| | 6.6. | ANALYSIS OF CI ENDPOINTS | 25 |

| | 6.7. | ADDITIONAL ANALYSIS | 26 |
|---|---|---|---|
| | | 6.7.1. ASES Comparison | |
| | | 6.7.3. Reoperation Surgery | |
| | | 6.7.4. ASES Shoulder Score – Within subject changes by visit | 29 |
| 7. | Table T | Cemplates (Tables, Figures, Listings - TFL) | 30 |
| | 7.1. | FREQUENCIES | 30 |
| | 7.2. | DESCRIPTIVE STATISTICS | 30 |
| | 7.3. | LISTINGS | 31 |
| 8. | Referen | 1CPS | 32 |

# 1. Administrative Information

### 1.1. LIST OF ABBREVIATIONS

| <u>Acronym</u> | <u>Definition</u> |
|----------------|--------------------------------------|
| ADE | Adverse Device Event |
| AE | Adverse Event |
| ASES | American Shoulder and Elbow Surgeons |
| CI | Confidence Interval |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| FR | Final Report |
| ICF | Informed Consent Form |
| IFU | Instructions for Use |
| IR | Interim/Annual Report |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| LTFU | Lost to Follow-Up |
| PP | Per Protocol |
| RSA | Reverse Shoulder Arthroplasty |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| TFL | Tables, Figures, Listings |
| TSA | Total Shoulder Arthroplasty |
| UADE | Unanticipated Adverse Device Effect |

### 1.2. STATISTICAL ANALYSIS PLAN REVISION HISTORY

| Version | Effective Date | Description | Reason |
|---------|----------------|-----------------|---------------------|
| 1 | 27OCT2020 | Initial Version | |
| 2 | 2 28MAY2021 | | Revision DQI 20-048 |

#### 1.3. ROLES AND RESPONSIBILITIES

| Role | Contributor | Affiliation |
|--------------------------------------|-----------------|-------------|
| Author | Sascha Lorenzen | Stryker |
| (Senior) Statistician | Claudia Beimel | Stryker |
| Clinical Research Head (CRH) | Rebecca Gibson | Stryker |
| Clinical Investigation Manager (CIM) | Susanne Höfer | Stryker |

### 2. Introduction

#### 2.1. BACKGROUND AND RATIONALE

The ReUnion TSA System is designed as an anatomical total shoulder or hemi-shoulder endoprosthesis to address advanced arthritic disorders affecting the shoulder joint in subjects having intact or repairable rotator cuff function. The ReUnion TSA System consists of a completely modular shoulder platform including a Humeral Stem, Humeral Head and Glenoid. The intended purposes of the ReUnion TSA System are to achieve pain relief, improvement of range of motion and restoration or improvement of the shoulder function while ensuring long-term replacement of the shoulder joint with sufficient stability of all endoprosthesis components.

#### 2.2. CLINICAL INVESTIGATION DESIGN

This investigation is a prospective, multicenter clinical investigation. It is anticipated that a total of one hundred (100) subjects will be enrolled at approximately 4-7 sites. Neither subjects nor investigators are blinded to treatment and the clinical investigation does not include a contemporaneous control. The clinical investigation has been designed to follow the surgeon's standard of care for shoulder arthroplasty subjects, which entails clinical evaluation on a regular ongoing basis, or as needed should the subject become symptomatic in the treated joint. The enrollment period is expected to occur over 14 months.

### 3. Research Goals

#### 3.1. FRAMEWORK

All quantitative variables, including those based on calculations (secondary elements), will be analyzed with a case summary evaluation before the detailed characteristics and parameters can be evaluated. A case summary contains a listing of the number of valid cases/values, missing cases/values (if any) and total cases/values in the specific analysis. In general, a central position parameter for quantitative variables the mean, median and mode will be analyzed. As variation parameter the standard deviation, 95% confidence interval of the mean, interquartile range and range (based on maximum and minimum) will be calculated. All quantitative variables will be assessed for normality using the Shapiro-Wilk test. For optional visualization of quantitative variables, box-and-whisker plots will be used. Additional analyses like skewness and kurtosis measures or standard errors are optional also.

All qualitative variables, including those based on summaries (secondary elements), will be analyzed listing the proportions, frequencies, column and row totals, and missing proportion (if any).

### 3.1.1. Primary Analysis / Endpoint

The objective of the clinical investigation is to demonstrate non-inferiority (equal or better) of the ASES Shoulder Score in relationship to the officially cleared indications in comparison to respective clinical outcome data in the scientific literature.

Data collection of ASES Shoulder Score will start pre-operatively and will be collected according to schedule in Table 4.4 This will be repeated annually in all subjects who have the total or partial prosthesis with full or partial implant survival (including all subjects without removal of all endo-prosthesis components).

The 24 months postoperative results for subjects implanted with ReUnion TSA System will be compared to a historical group and results reported by respective clinical outcome data in the scientific literature. The benchmark sources and values will serve as the control group for the ReUnion TSA System subjects.

Higher ASES Shoulder Score results are linked to better subject results and vice versa.

The clinical investigation endpoint is non-inferiority to the control, meaning the clinical investigation result should be equal or better than the control. In this clinical investigation, an equal or better ASES Shoulder Score result means equal or more  $(\ge)$ . As only results from samples will be captured, results mostly are estimates of the true population parameter. These estimates vary by a certain area, where it is expected that the true population parameter falls within. Based on this, it is required to specify a lower limit for the acceptable difference or zone of indifference, denoted as  $-\theta$ .

Hypotheses were developed to allow for a comparison of the 24 months postoperative ASES Shoulder Score effectiveness / performance between the two underlying populations. The 24 months postoperative ASES Shoulder Score is the primary endpoint of this clinical investigation. Hypothesis tests will be one-sided with a significance level  $\alpha$  of 5%.

| Hypothesis Eq | uations | Interpretation |
|---|---|---|
| Null (H0) | $A - B < -\theta$ | Central tendency of A is inferior to the |
| | ReUnion TSA Syste<br>Control (Benchmark | |
| Alternative (H1) | $A - B \ge -\theta$ | Central tendency of A is non-inferior to |
| 7 Hermanye (111) | ReUnion TSA Syste<br>Control (Benchmark | |
| | - θ | 95%<br>H <sub>1</sub> |
| Possible<br>Evidence (p) | Possible<br>Decisions | Possible Conclusions – ASES Shoulder Score |

| p-value > α (0.05) | Fail to reject<br>null hypothesis<br>(H0) | ReUnion TSA System < Control (Benchmark)<br>Insufficient evidence to reject the null hypothesis<br>(H0: A - B < - $\theta$ ) at the pre-determined significance<br>level of 5%. |
|---|---|---|
| p-value $\leq \alpha (0.05)$ | Reject null<br>hypothesis (H1) | ReUnion TSA System $\geq$ Control (Benchmark)<br>Sufficient evidence to reject the null hypothesis<br>(H0: A - B < - $\theta$ ) at the pre-determined significance<br>level of 5%. |

Table 3.1.1: Research Goal and Hypothesis (Primary Endpoint)

To test non-inferiority, the 24 months mean ASES Shoulder Score result of the ReUnion TSA System group will be compared to the mean estimate of the control group, 82.16 points.

To be able to identify an acceptable difference or zone of indifference  $(-\theta)$ , the pooled standard deviation of the ASES Shoulder Score result at 24 months postoperative in the control group (Benchmark) was used as lower limit (pooled standard deviation of control is 16.76 points). The lower maximum acceptable difference  $(-\theta)$  is 65.40 points (mean of control -  $\theta$  or 82.16 – 16.76 = 65.40 points).

Based on the underlying distribution of the data and the result of the normality assessment, either the parametric one-sample t-test or the non-parametric one-sample sign test will be used to compare the 24 months postoperative ASES Shoulder Score results of the ReUnion TSA System against the value of 65.40 points.

The analysis of the primary endpoint / objective will be conducted when all subjects have completed the 24 months postoperative including the ASES Shoulder Score.

### 3.1.2. Secondary Analyses

For safety, the incidence of device-related adverse events/incidents will be assessed up to 10 years after the index procedure and monitored through collection and analyses.

Furthermore, time to (earliest) Device-Related Adverse Events will be analyzed as well. For analysis of the time to the (earliest) Device-Related Adverse Events, the Kaplan-Meier method will be used. Considered variables, the level of measurement and the planned analysis steps are listed in detail in the SAP. These analyses will be part of the final report.

#### 3.1.3. Additional Analyses

Additional Analyses are outlined in the subsequent sections. Analysis details (variables, level of measurement, planned steps) are listed in-depth in the SAP.

#### o Mortality

For analysis of the time to death or mortality, the Kaplan-Meier method will be used. The times between surgery and the last available assessment will be used together with the times between date of surgery and the date of death. This analysis will be part of the final report.

### • ASES Total Score – Within subject changes by visit

The within subject score changes of the ASES Total Score from visit to visit will be analyzed to help identify the changes on the subject level. This analysis will be part of the final report.

#### 3.2. SAMPLE SIZE

The determination of sample size is based on benchmark sources and values. To account for an estimated appropriate overall drop-out rate, Stryker intends to enroll the calculated number of subjects, multiplied

by the number of cleared indications to reflect the underlying subject population adequately. For details, please see Table 3.2.

| Benchi | mark and Objective | es for Cli | nical Inve | estigation | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Endpo | int | Non-inferiority (equal or better) of the ASES Shoulder Score in relationship to the officially cleared indications in comparison to respective clinical outcome data in the scientific literature. | | | | | | | |
| | | 56% (co | nfirmed l | y Medica | ıl Expert, | see Cuff | et al.) | | |
| Estimated drop-out rate Cuff et al. Reverse Shoulder Arthroplasty for the Treatment of Rot Deficiency: A Concise Follow-up, at a Minimum of 10 Years, of F Reports. J Bone Joint Surg Am. 2017 Nov 15;99(22):1895-1899. 10.2106/JBJS.17.00175. | | | | | | Previous | | | |
| Benchi | mark Sources & Va | lues ASE | S [points | ] | | | | | |
| Source | ; | | n | Mean | Std.<br>Dev. | | С | omments<br>No. | |
| No. | Title | | | | | | | | |
| 1 | Irlenbusch et al. [3 | 10] | 73 | 77.9 | N/A | | stract vs r | d to Follo<br>nethod vs | w-Up times<br>result |
| 2 | Flurin et al. [20] | | 73 | 90.3 | 14.6 | Not c | lear if SE | or 95% ( | CI |
| 3 | Press et al. [22] | 34 | 82.6 | 19.4 | | | | | |
| 4 | Hsu et al. [23] | | 25 | 94.4 | N/A | | | | |
| 5 | Kiet et al. [26] | | 40 | 80 | 21 | | | m 45 to 40 | |
| 6 | Steen et al. [29] | | 96 | 80.4 | 22.4 | Not c | Not clear if SD or 95% CI | | |
| 7 | Gulotta et al. [34] | | 40 | 80.1 | 10.1 | | | | |
| 8 | Petri et al. [49] | Petri et al. [49] | | | 13.1 | | | | |
| 9 | Schoch et al. [62] | | 78 | 88.4 | 16.7 | | | | |
| 10 | Alentorn-Geli et a | 1. [70] | 38 | 64 | N/A | TSA | TSA und HA combined. | | |
| Identif | fied Cleared Indicat | ions | | | | | | | |
| No. | Indication | | | | | | | | |
| 1 | Post-traumatic art | hritis | | | | | | | |
| 2 | Degenerative arth | | | | | | | | |
| 3 | Rheumatoid arthri | | | | | | | | |
| 4 | Revision of previo | ously faile | ed shoulde | er joint rep | lacement | : | | | - |
| 5 | Aseptic necrosis | | | | | | | | |
| Explor | ative Meta-Analysi | is - ASES | (single g | roup) | | | | | |
| Accept | tance Criteria | | | | | | | | |
| Confid | lence Interval (CI) | | | | | 0.95 ( | (95%) tw | o-sided | |
| Softwa | re Used | | | | | IBM | SPSS V2 | 0 | |
| | | | Case I | Processing S | Summary | ı | | | |
| | | | | | Cas | es | | | |
| | | | Va | lid | Miss | ing | ing Tot | | |
| | | | N | Percent | N | Percent | N | Percent | |
| | Mean ASES ReUnion_TSA_CE | R | 10 | 100,0% | 0 | 0,0% | 10 | 100,0% | |
| | Std.Dev. ASES<br>ReUnion_TSA_CE | R | 7 | 70,0% | 3 | 30,0% | 10 | 100,0% | |

| Descriptives | | | |
|-----------------|-------------------------|-------------|-----------|
| | | | Statistic |
| Std.Dev. ASES | Mean | | 16,7571 |
| ReUnion_TSA_CER | 95% Confidence Interval | Lower Bound | 12,6353 |
| | for Mean | Upper Bound | 20,8790 |
| | Median | | 16,7000 |
| | Std. Deviation | | 4,45678 |
| | Minimum | Minimum | |
| | Maximum | Maximum | |
| | Interquartile Range | | 7,90 |
| Mean ASES | Mean | | 82,1600 |
| ReUnion_TSA_CER | 95% Confidence Interval | Lower Bound | 76,2372 |
| | for Mean | Upper Bound | 88,0828 |
| | Median | | 81,5000 |
| | Std. Deviation | | 8,27945 |
| | Minimum | | 64,00 |
| | Maximum | | 94,40 |
| | Interquartile Range | | 9,40 |



Red line: Pooled mean ASES Blue lines: 95% CI of pooled mean

**ASES** 

Black line: Pooled median pooled

**ASES** 

Box: Interquartile Range

Green Line: Pooled mean ASES minus pooled std. dev. ASES

(16.76)

82.16 - 16.76 = 65.40 points

| Acceptance Criteria for Sample Size Calculation | | |
|---|---|---|
| Significance Level (α) | 0.05 (5%) | |
| Power (1-β) | 0.80 (80%) | |
| Confidence Interval (CI) | 0.95 (95%) | |
| Tails | 2 | |
| Path | Non-inferiority – ReUnion TSA (A) $\geq$ Benchmark (B, explorative meta-analysis in this document) | |
| Hymotheses Poin | Null (H <sub>0</sub> ) | $A - B < -\theta$ |
| Hypotheses Pair | Alternative (H <sub>1</sub> ) | $A - B \ge -\theta$ |
| Benchmark Timepoint | 24 months postoperative | |
| Benchmark n (sources) | 10 | |
| Benchmark Mean | 82.16 (pooled mean ASES [points]) | |
| Benchmark Std. Dev. | 16.76 (pooled std. dev. ASES [points]) | |
| Benchmark Value<br>Non-Inferiority Margin (-θ) | Pooled mean ASES minus pooled std. dev. ASES (16.76) 82.16 – 16.76 = <b>65.40 points</b> | |
| Software Used | IBM SPSS Sample Power V3.0 | |

### **IBM SPSS Sample Power Output**

One goal of the proposed clinical investigation is to test the null hypothesis that the population mean is 82.16 points. The criterion for significance (alpha) has been set at 0.05. The test is 2-tailed, which means that effects in both directions will be interpreted. With the proposed sample size of 10 cases, the clinical investigation will have power of 80.3% to yield a statistically significant result. This computation assumes

that the population from which the sample will be drawn has a mean of 82.16 points with a standard deviation of 16.76 points. The observed value will be tested against a theoretical value (constant, noninferiority margin) of 65.40 points. IBM SPSS Sample Power Output - Screenshot IBM SPSS SamplePower - [ One-sample t-test] П × <u>File View Options Tools Scenarios Help</u> \_ B × 95% Population Mean Standard 95% Standard N of Cases Deviation Lower Upper Expected mean 10 82,16 16,76 5,30 70,62 93.70 Test against the constant 65,40 Alpha= 0,050, Tails= 2 Power = 0,803 Estimated overall drop-out rate is 56% which leads to the requirement of enrolling additional 6 subjects into the clinical investigation. Number of subjects to be enrolled: 16 subjects Sample Size (rounded up to 20 subjects) Overall Sample Size (multiplied by 100 subjects number of indications (=5)

Table 3.2: Sample Size Justification

In conclusion, the calculated number of subjects to be enrolled (10), plus the estimated overall drop-out rate of 56%, leads Stryker's enroll 20 subjects per cleared indication (5) to reflect the underlying subject population adequately. As a result, an enrollment target of 100 subjects in total will be aspired (ideally, but not necessarily, composed with 20 subjects per indication).

### 4. Methods

#### 4.1. RANDOMIZATION

No specific methods for assigning subjects will be used for this clinical investigation. A consecutive series of subjects at each site meeting all the eligibility criteria will be enrolled in this clinical investigation.

#### 4.2. STATISTICAL INTERIM ANALYSES AND STOPPING GUIDANCE

Interim analyses will be performed on a yearly basis. The progress of the clinical investigation will be reported together with the interim results on the variable level according to the analysis plan.

The analysis of the primary endpoint / objective will be part of the related interim / annual report when all subjects have completed the 24 months postoperative including the ASES Shoulder Score.

There will be no stopping rules specified for this clinical investigation.

#### 4.3. TIMING OF FINAL ANALYSES

The full final report with complete analysis, progress and conduct reporting will be created at the end of this clinical investigation.

#### 4.4. TIMING OF OUTCOME ASSESSMENT

Subjects in this clinical investigation will be evaluated at Pre-Operative, Operative/Discharge, and at 6 Weeks (4 weeks – 8 weeks), 6 Months (24 weeks – 28 weeks), 12 Months (48 weeks- 56 weeks), 24

Months (100 weeks – 108 weeks) and annually after the index procedure. The follow-up evaluations will include assessment of device-related AEs/incidents, radiographs and ASES Shoulder Score.

| Assessment | | | Preoperative | Operative/<br>Discharge | 6 Weeks <sup>a, b</sup> (+/- 2 weeks) | 6 Months <sup>a, b</sup> (+/- 3weeks) | 12 Months <sup>a, b</sup> (+/- 4 weeks) | 24 Months <sup>a, b</sup> (+/- 4 weeks) | Annually <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Informed Conse | ent | | X | | | | | | |
| Demographics of | | edical History | X | | | | | | |
| Inclusion/Exclu | ısion | | X | | | | | | |
| Physical Exam | | | X | | Xc | Xc | Xc | Xc | Xc |
| Surgical Proced | | | X | X | | | | | |
| | ASES Shoulder Score | | | | Xd | X <sup>d</sup> | X <sup>d</sup> | Xd | X <sup>d</sup> |
| Image Evaluation e, f | | X | X | X | X | X | X | X | |
| Subject Disposition <sup>g</sup> | | | | X | X | X | X | X | |
| Device-Related AEs/ | | | ncidents & | z Reoperati | ons will be | collected t | throughout | the course | of the |
| | a. | Follow-up visit so | chedule to | reflect Inst | itutions' St | andard of C | Care praction | ces | |
| b. If the subject mis made to collect d | | | | | | | v, then eve | ry effort sl | ould be |
| | c. Evaluation may be collected when subject presents in-clinic for study visit. | | | | | | | | |
| d. Evaluation can be | | | collected | via phone. | | | | | |
| | | | ection should follow Institution's Standard of Care practices and no should be made for study purposes. | | | | | | |
| f. CT scans may be collected if part of Institution's Standard of Care practices. | | | | | | | | | |
| | g. | Subject Disposition to the completion | | | | time point | for subject | withdrawa | l prior |

Table 4.4: Schedule of Events

#### 4.5. STATISTICAL SOFTWARE

Statistical Analysis will be performed using IBM SPSS, IBM SPSS Sample Power as well as established standard software packages (e.g. MS Excel).

#### 4.6. MISSING DATA

The intent is to collect as complete a dataset as possible. Nevertheless, in some situations missing data cannot be avoided. The reports and tables therefore will show the number and percentage of missing cases for each analyzed variable in relation to the enrolled cases for each postoperative assessment

Any deviations from Statistical Analysis Plan will be listed in the annual or final reports.

### 4.7. CONFIDENCE INTERVALS AND P-VALUES

The following acceptance / rejection criteria were used for this clinical investigation:

| Parameter | Acceptance / rejection criteria |
|---------------------------------|---------------------------------|
| Confidence level (1-α) | 0.95 (95%) |
| Significance level (α) | 0.05 (5%) |
| Power (1-β) | 0.80 (80%) |
| Beta-level (β) | 0.20 (20%) |
| Confidence interval of mean | 95% |
| p-value indicating significance | ≤ 0.05 |

Table 4.7: Acceptance / Rejection Criteria

#### 4.8. UNITS

See analysis chapter for details related to units used for the different variables and calculations.

In case of collection of variables with non-SI units (e.g. pounds instead to kilograms), conversion of such data into SI units (and vice versa) will be ensured and both results will be reported for the full set of available subjects next to each other in the interim/annual and/or final reports.

#### 4.9. CALCULATIONS AND TRANSFORMATIONS

Distances between times and differences between score results will be calculated. For full details of variables used for calculations and the creation of new variables based on these calculations, see analysis chapter.

#### 4.10. ASSUMTIONS

In case of deviation from assumptions (e.g. normality), non-parametric methods will be used for analysis. No transformation of such data will be performed.

### 5. Population and Progress

#### 5.1. ANALYSIS POPULATION

It is expected that during this clinical investigation only one population for ReUnion TSA System will exist and all subjects will be analyzed "Per Protocol" (PP). However, it cannot be fully avoided that in theory subjects might need to be excluded from the PP population. In this occasion, there will be two groups being fully analyzed to ensure transparency and avoid bias.

The groups are defined as follows:

### • Intent-to Treat Population

The Intent-to-Treat (ITT) Population is defined to be all enrolled subjects. An enrolled subject is a subject that has signed informed consent, all screening procedures have been successfully completed, is eligible and can receive treatment. The ITT population will not be analyzed for the annual reports and will only be included in the final report.

#### • Per Protocol Population

The PP Population is defined to be all subjects in the ITT Population with no major CIP violations. The CIP violations that will exclude a subject are as follows:

- The subject does not receive the ReUnion TSA System
- The subject does not meet all eligibility criteria
- The subject has a clinical investigation plan violation that is considered likely to affect subject outcomes.

After the clinical investigation has been completed, a review of the data will be conducted to determine which subjects are to be excluded from the PP population.

The following tables will be created for interim/annual and final reports related to the clinical investigation populations and progress:

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan |
|---|---|---|
| All Forms - Overview & Progre | ss Report | |
| Counting of available subjects <b>Subject Population by Site</b> (Variable(s): SITENUM; SUBID) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of available subjects Subject Population by Visit (Variable(s): SITENUM; SUBID; VISITDT) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of available subjects Subject Population by Visit and by Site (Variable(s): SITENUM; SUBID; VISITDT) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |

Table 5.1: Populations and Progress Tables List

#### 5.2. ELIGIBILITY

A subject is defined as eligible if all inclusion and exclusion criteria are fulfilled as it is described in the clinical investigation plan. For details see CIP.

For tables to be created for the interim/annual and final reports, see chapter 6.2 and tables list 6.2.2.

#### 5.3. WITHDRAWAL/FOLLOW-UP

During the clinical investigation if a subject must be withdrawn prematurely from the clinical investigation, then the procedures outlined in the CIP should be followed. These procedures should not interfere with the initiation of any new treatments that are necessary to treat a subject's condition. Information on all withdrawn subjects will be documented.

The following tables will be created for interim/annual and final reports related to the numbers of withdrawn subjects (if any):

| Evaluation | Level of | Analysis Plan |
|---|---|---|
| Variable / Question | Measurement | Analysis I lan |
| All Forms - Overview & Progre | ss Report | |
| Counting of withdrawn subjects Number of Subjects Withdrawn by Site (Variable(s): SITENUM; COMPPROT; PRIMRSN) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Counting of withdrawn subjects Number of Subjects Withdrawn by Site by Visit (Variable(s): SITENUM; COMPPROT; PRIMRSN; VISITDT) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). |
| Comments related to Reasons for<br>Subjects Withdrawn<br>(Variable(s): RSNSPF) | Text, String | Listing of reasons for subjects being excluded by subject code/ID |

Table 5.3: Withdrawal Tables List

### 5.4. ADHERENCE AND CIP DEVIATIONS

Any CIP deviations will be listed in the interim/annual and final reports. It is optional to describe this chapter in free text or present it in a tabulated format.

# 6. Analysis

The following tabulated analysis plan reflects this approach and specifies the variables characteristics (quantitative or qualitative) in detail together with the related analysis strategy. This also includes calculation and summaries based on primary elements and the required analysis.

In addition, it will be defined in the text or directly in the tables below, if the variable must be included in an interim/annual report (IR) and/or in the final report (FR).

### 6.1. HARMS AND SAFETY

Categorization and definitions of (Serious-, Unanticipated-) Adverse Device Effects, (Serious-) Incidents are given in the CIP.

The following tables will be created for interim/annual and final reports related harms and safety:

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | I | Inclusion | |
|---|---|---|---|---|---|
| Adverse Events / Incidents | | | IR | FR | N/A |
| Perioperative/Postoperative AE<br>(Variable(s): PERPOST) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Device-Related Adverse Event /<br>Incident<br>(Variable(s): AEEVENT; AEOTHER) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of other Events/Incidents. | X | X | |
| Describe the AE/Incident<br>(Variable(s): AEDESCRP) | Qualitative, nominal | Listing of other<br>Events/Incidents Description. | | | X |
| Unanticipated Adverse Device<br>Event?<br>(Variable(s): AEUADE) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Severity<br>(Variable(s): AESEVER) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Action Taken<br>(Variable(s): ACTNONE; ACTMEDS;<br>ACTSURG; ACTSHORT;<br>ACTPROHS; ACTOTHER;<br>ACTOTHSP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given Other specifications. | | | X |
| AE Resolution<br>(Variable(s): AERESOLV) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Outcome<br>(Variable(s): AEONWOTR;<br>AEONWTTR; AEREWOTR;<br>AEREWTTR; AETEDISB;<br>AEPERMD; AESUEXP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Creation of variable Number of Adverse Device Effects by Site (Variable(s): AEEVENT; SITENUM) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Creation of variable Number of<br>Adverse Device Effects per Subject<br>and Site<br>(Variable(s): AEEVENT; SITENUM;<br>SUBID) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |

Table 6.1.1: Adverse Events / Incidents Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | n |
|---|---|---|---|---|---|
| Reoperation | | | IR | FR | N/A |
| Type of Procedure (Variable(s): IRRDEB; SOFTTR; ROTCUFF; OTHSOFT; REVHATSA; REVHATSASP; CONTSAWHS; CONTSAWOHS; CONRSAWHS; CONRSAWOHS; CONHAWHS; CONHAWOHS; CONTRSAWHS; CONTRSAWOHS; REVINFEC; REVINFECSP; RESSALV; ARTHSJ; ORIF; RESOST; PTOTHR; PTOTHSPC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listings of implant specifications. | X | X | |
| Reason(s) for Reoperation (Variable(s): WOUNCOM; INFEC; NERPL; DISLOC; OTHSUB; MALIMP; UNDOV; IMPDISL; ROTCUFTR; EROSHA; IMPLOOS; IMPBRKG; WRGLENTSA; PERIFRAC; STIFF; PAIN; HETOSS; RROTH; RROTHSP) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listings of other specifications. | X | X | |

Table 6.1.2: Reoperation Tables List

### 6.2. BASELINE CHARACTERISTICS

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | n |
|---|---|---|---|---|
| Preoperative Visit Form – Subject Eligibility – Inclusion & Exclusion Criteria | | | | N/A |
| Note: Inclusion and exclusion criteria will be checked during monitoring and reported by a statement (e.g. all subjects fulfilled the inclusion criteria). | | | | |
| Inclusion Criteria Questions<br>(Variable(s): INCLA; INCLB; INCLC;<br>INCLD) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Exclusion Criteria Questions<br>(Variable(s): EXCLA; EXCLB;<br>EXCLC; EXCLD; EXCLE; EXCLF;<br>EXCLG; EXCLH) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Creation of variable No. of Eligible Subjects. Conclusion of Inclusion and Exclusion Questions. | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |

Table 6.2.1: Preoperative Visit Form - Subject Eligibility – Inclusion & Exclusion Criteria
Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | n |
|---|---|---|---|---|---|
| Preoperative Visit Form - Subje | ect Demographic | s | IR | FR | N/A |
| Creation of variable Age [years] Difference between Date of Surgery [dd.mmm.yyyy] and Date of Birth/DOB [dd.mmm.yyyy] in [ years ] (Variable(s): BIRTHDT; VISITDT; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| Gender<br>(Variable(s): GENDER) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Race (Variable(s): AMERIND; ASIAN; BLKAFR; NATHAW; CAUS; RACEOTH; RACEOTHR) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |

| | | Listing of given specifications. | | | |
|---|---|---|---|---|---|
| Height [captured in inches or cm] In the analysis, all values will be reported in inches and cm next to each other. (Variable(s): HGHTM) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | X |
| Weight [captured in lbs or kg] In the analysis, all values will be reported in lbs and kg next to each other. (Variable(s): WEIGHTKG) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | X |
| Body Mass Index [kg/m²]<br>(Variable(s): BMI) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |

Table 6.2.2: Preoperative Visit Form - Subject Demographics Tables List

| Evaluation Variable / Question Preoperative Visit Form – Curr | Level of<br>Measurement<br>ent Relevant Me | Analysis Plan | In<br>IR | nclusio<br>FR | n<br>N/A |
|---|---|---|---|---|---|
| Current Relevant Medical<br>Conditions (Variable(s): CURCOND;<br>CONDSPC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |

Table 6.2.3: Preoperative Visit Form - Current Relevant Medical Conditions

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Iı | nclusio | n |
|---|---|---|---|---|---|
| Preoperative Visit Form - Subjection | ect Evaluation | | IR | FR | N/A |
| Tobacco Use:<br>(Variable(s): TOBCCO) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Corticosteroids Taking:<br>(Variable(s): CORTICO) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Affected (Study) Shoulder<br>(Variable(s): AFFCSHL) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Primary Shoulder Diagnosis:<br>(Variable(s): PRIMDIAG) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | X | |
| Shoulder Arthroplasty Procedure:<br>(Variable(s): SHLARPROC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given specifications. | X | X | |
| Previous History of Surgery to the<br>Affected Shoulder<br>(Variable(s): PREVHIST) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |

| | | Listing of given specifications. | |
|---|---|---|---|
| Procedure 1<br>(Variable(s): PROCNM1) | Text, String | Listing of comments and | X |
| Procedure Date 1<br>(Variable(s): PROCDT1) | Quantitative, ratio Date/Time | dates together identified by subject code/ID | X |
| Procedure 2<br>(Variable(s): PROCNM2) | Text, String | Listing of comments and | X |
| Procedure Date 2<br>(Variable(s): PROCDT2) | Quantitative, ratio Date/Time | dates together identified by subject code/ID | X |
| Procedure 3<br>(Variable(s): PROCNM3) | Text, String | Listing of comments and | X |
| Procedure Date 3<br>(Variable(s): PROCDT3) | Quantitative, ratio Date/Time | dates together identified by subject code/ID | X |
| Procedure 4<br>(Variable(s): PROCNM4) | Text, String | Listing of comments and | X |
| Procedure Date 4<br>(Variable(s): PROCDT4) | Quantitative, ratio Date/Time | dates together identified by subject code/ID | X |

Table 6.2.4: Preoperative Visit Form – Medical History Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | on |
|---|---|---|---|---|---|
| Preoperative Visit Form – ASE | | e (prior to surgery) | IR | FR | N/A |
| Q1 - Usual Work<br>(Variable(s): USWORK) | Text, String | Listing of comments identified by subject code/ID | | | X |
| Q2 - Usual Sport/Leisure activity?<br>(Variable(s): USSPRT) | Text, String | Listing of comments identified by subject code/ID | | | X |
| Q3 - Do you have shoulder pain at night? (Variable(s): PNNIGHT) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q4 - Do you take pain killers such as<br>paracetamol (acetaminophen),<br>diclofenac, or ibuprofen?<br>(Variable(s): PNKLR) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q5 - Do you take strong pain killers<br>such as codeine, tramadol, or<br>morphine?<br>(Variable(s): CODTRMD) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q6 - How many pills do you take on<br>an average day?<br>(Variable(s): PILLNUM) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | X |
| Q7 - Intensity of pain? (Variable(s): PAINC) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | | X |
| Q8 - Is it difficult for you to put on a coat? (Variable(s): PUTCOAT) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |

| 00 7 1 1100 1:0 | T | I B | | | 1 |
|---|---|---|---|---|---|
| Q9 - Is it difficult for you to sleep on the affected side? | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, | | | X |
| (Variable(s): DIFSLP) Q10 - Is it difficult for you to wash | Qualitative, | missing proportion (if any). Proportions, frequencies, | | | |
| your back/do up bra?<br>(Variable(s): WASHBCK) | Ordinal | column and row totals, missing proportion (if any). | | | X |
| Q11 - Is it difficult for you manage toileting? | Qualitative, | Proportions, frequencies, column and row totals, | | | Х |
| (Variable(s): MNGTOIL) | Ordinal | missing proportion (if any). | | | Λ |
| Q12 - Is it difficult for you to comb<br>your hair?<br>(Variable(s): COMBHR) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q13 - Is it difficult for you to reach a high shelf? (Variable(s): HIGHSHL) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q14 - Is it difficult for you to lift<br>10lbs. (4.5kg) above your shoulder?<br>(Variable(s): LIFT10) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q15 - Is it difficult for you to throw a ball overhand?<br>(Variable(s): BALLOV) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q16 - Is it difficult for you to do your usual work? (Variable(s): DFWORK) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| Q17 - Is it difficult for you to do your usual sport/leisure activity? (Variable(s): SPRACT) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | | X |
| ASES Pain Score [points] (Variable(s): PAINSC) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |
| ASES Functioning Score [points] (Variable(s): FUNSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | Х | Х | |
| Total ASES Shoulder Score [points] (Variable(s): FINSCORE) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | X | X | |

Table 6.2.5: Preoperative Visit Form – ASES Shoulder Score (post fracture, prior to surgery) Tables

List

### 6.3. INTRAOPERATIVE CHARACTERISTICS

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusio | | n |
|---|---|---|---|---|---|
| Operative Visit – Operative Pro | | | IR | FR | N/A |
| Date of Surgery [dd.mmm.yyyy]: (Variable(s): VISITDT; VISNAME) | Date/Time | Listing the first and last surgery in the report text to describe from which date to which date subjects were operated. | | X | |
| Date of Admission [dd.mmm.yyyy]:<br>(Variable(s): ADMINDT) | Date/Time | None | | | X |
| <b>Date of Discharge </b> [dd.mmm.yyyy]: (Variable(s): DISCHRDT) | Date/Time | None | | | X |
| Creation of variable Difference between Date of Surgery [dd.mmm.yyyy] and Date of Discharge [dd.mmm.yyyy] in [ days J (Variable(s): VISITDT; DISCHRDT; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Surgery Start Time (24-hour clock): (Variable(s): SURGSTTM) | Date/Time | None | | | X |
| Surgery Stop Time (24-hour clock): (Variable(s): SURGSPTM) | Date/Time | None | | | X |
| Difference between Surgery Start Time and Surgery Stop Time in [ hh:mm ] (Variable(s): SURGSTTM; SURGSPTM) | Quantitative,<br>ratio<br>Date/Time | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Amount of Blood Infused<br>(Variable(s): BLOODINF) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Type of Anesthesia:<br>(Variable(s): TYPANEST) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Were there any technical difficulties<br>during surgery?<br>(Variable(s): SURGDIFF;<br>SURGDESC) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | X | X | |
| Were any concomitant procedures<br>done during surgery?<br>(Variable(s): CONPROC;<br>CONPROCD) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | X | X | |

Table 6.3.1: Operative Visit – Surgical Procedure Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | |
|---|---|---|---|---|---|
| Operative Visit – Implant Specification | | | IR | FR | N/A |
| Humeral Stem Lot/Serial # (Variable(s): HSREF) | Qualitative,<br>nominal | None, used to populate diameter, length, press-fit | | X | |

| | | textured or smooth uncoated stem details Proportions, frequencies, column and row totals, missing proportion (if any). | |
|---|---|---|---|
| Humeral Head Lot/Serial # (Variable(s): HHREF) | Qualitative,<br>nominal | None, used to populate diameter, thickness and standard(eccentric humeral head details Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Glenoid Lot/Serial #<br>(Variable(s): GLENREF) | Qualitative,<br>nominal | None, used to populate size<br>and pegged/keeled glenoid<br>details<br>Proportions, frequencies,<br>column and row totals,<br>missing proportion (if any). | х |

Table 6.3.2: Operative Visit – Implant Specification Tables List

| Evaluation | Level of | Analysis Plan | Inclusion | | |
|---|---|---|---|---|---|
| Variable / Question | Measurement | Analysis I lan | liiciusioi | | -11 |
| Operative Visit - Radiographic | Evaluation | | IR | FR | N/A |
| Correct initial positioning of the | Qualitative, | Proportions, frequencies, | | | |
| humeral stem and head | nominal | column and row totals, | | X | |
| (Variable(s): QA) | | missing proportion (if any). | | | |
| Correct sizing of the humeral stem | Qualitative, | Proportions, frequencies, | | | |
| and | nominal | column and row totals, | | X | |
| head | | missing proportion (if any). | | 71 | |
| (Variable(s): QB) | | | | | |
| Correct positioning of the glenoid | Qualitative, | Proportions, frequencies, | | | |
| component | nominal | column and row totals, | X | | |
| (Variable(s): QC) | Homman | missing proportion (if any). | | | |
| Radiologic signs of intraoperative | Qualitative, | Proportions, frequencies, | | | |
| fracture of the humerus | nominal | column and row totals, | X | | |
| (Variable(s): QD) | Homman | missing proportion (if any). | | | |
| Radiologic signs of intraoperative | nominal c | Proportions, frequencies, | | | |
| fracture of the glenoid | | column and row totals, | | X | |
| (Variable(s): QE) | | missing proportion (if any). | | | |
| Correct cementation of the humeral | Qualitative, | Proportions, frequencies, | | | |
| component | nominal | column and row totals, | | X | |
| (Variable(s): QF) | Hommun | missing proportion (if any). | | | |
| Correct cementation of the glenoid | Qualitative, | Proportions, frequencies, | | | |
| component | nominal | column and row totals, | | X | |
| (Variable(s): QG) | Homman | missing proportion (if any). | | | |
| Radiologic signs of humeral cement | Qualitative, | Proportions, frequencies, | | | |
| leakage | nominal | column and row totals, | | X | |
| (Variable(s): QH) | Homman | missing proportion (if any). | | | |
| Radiologic signs of glenoidal cement | Qualitative, | Proportions, frequencies, | | | |
| leakage | nominal | column and row totals, | | X | |
| (Variable(s): QI) | | missing proportion (if any). | | | |
| Other | Qualitative, | Proportions, frequencies, | | | |
| (Variable(s): QJ) | nominal | column and row totals, | | X | |
| (, arraoto(s), Xs) | | missing proportion (if any). | 1 | | |
| Please describe the findings in detail | Qualitative, | Proportions, frequencies, | | | |
| (Variable(s): QDTL) | nominal | column and row totals, | | | X |
| ( · artaolo(b). QD1L) | | missing proportion (if any). | | | |

Table 6.3.3: Operative Visit Form – Radiographic Evaluation Tables List

# 6.4. EARLY POSTOPERATIVE CHARACTERISTICS

N/A

### 6.5. POSTOPERATIVE CHARACTERISTICS

The analysis of the Postoperative data must be performed separately for each follow-up visit listed in table 4.4 in accordance to the following tables in this chapter. New Variables must be created individually for each follow-up visit.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | n |
|---|---|---|---|---|---|
| Postoperative Visit Form – Date of Visit | | | | | N/A |
| Date of Visit [dd.mmm.yyyy]: | Date/Time | None | | | X |
| Creation of variable Difference between Date of Surgery [dd.mmm.yyyy] and Date of "FU Visit" [dd.mmm.yyyy] In [ days ] (Variable(s): VISITID; VISNAME) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | Х | |

Table 6.5.1: Postoperative Visit Form – Date of Visit

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | n |
|---|---|---|---|---|
| | Postoperative Visit Form – ASES Shoulder Score | | | N/A |
| Q1 - Usual Work<br>(Variable(s): USWORK) | Text, String | Listing of comments identified by subject code/ID | | X |
| Q2 - Usual Sport/Leisure activity?<br>(Variable(s): USSPRT) | Text, String | Listing of comments identified by subject code/ID | | X |
| Q3 - Do you have shoulder pain at night? (Variable(s): PNNIGHT) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Q4 - Do you take pain killers such as<br>paracetamol (acetaminophen),<br>diclofenac, or ibuprofen?<br>(Variable(s): PNKLR) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Q5 - Do you take strong pain killers<br>such as codeine, tramadol, or<br>morphine?<br>(Variable(s): CODTRMD) | Qualitative, nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |
| Q6 - How many pills do you take on<br>an average day?<br>(Variable(s): PILLNUM) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X |
| Q7 - Intensity of pain? (Variable(s): PAINC) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | Х |
| Q8 - Is it difficult for you to put on a coat? (Variable(s): PUTCOAT) | Qualitative,<br>Ordinal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X |

| 00 Is it different for your to also you | | Proportions, frequencies, | | | |
|---|---|---|---|---|---|
| Q9 - Is it difficult for you to sleep on the affected side? | Qualitative, | column and row totals, | | | X |
| (Variable(s): DIFSLP) | Ordinal | missing proportion (if any). | | | Λ |
| Q10 - Is it difficult for you to wash | | Proportions, frequencies, | | | |
| your back/do up bra? | Qualitative, | column and row totals, | | | X |
| (Variable(s): WASHBCK) | Ordinal | missing proportion (if any). | | | Λ |
| Q11 - Is it difficult for you manage | | Proportions, frequencies, | | | |
| toileting? | Qualitative, | column and row totals, | | | X |
| (Variable(s): MNGTOIL) | Ordinal | missing proportion (if any). | | | Λ |
| Q12 - Is it difficult for you to comb | | Proportions, frequencies, | | | |
| your hair? | Qualitative, | column and row totals, | | | X |
| (Variable(s): COMBHR) | Ordinal | missing proportion (if any). | | | Λ |
| Q13 - Is it difficult for you to reach a | | Proportions, frequencies, | | | |
| high shelf? | Qualitative, | column and row totals, | | | X |
| (Variable(s): HIGHSHL) | Ordinal | missing proportion (if any). | | | Λ |
| Q14 - Is it difficult for you to lift | Qualitative, | Proportions, frequencies, column and row totals, | | | 37 |
| 10lbs. (4.5kg) above your shoulder? | Ordinal | | | | X |
| (Variable(s): LIFT10) | | missing proportion (if any). | - | | |
| Q15 - Is it difficult for you to throw a | Qualitative, | Proportions, frequencies, | | | 37 |
| ball overhand? | Ordinal | column and row totals, | | | X |
| (Variable(s): BALLOV) | | missing proportion (if any). | | | |
| Q16 - Is it difficult for you to do your | Qualitative, | Proportions, frequencies, | | | |
| usual work? | Ordinal | column and row totals, | | | X |
| (Variable(s): DFWORK) | | missing proportion (if any). | | | |
| Q17 - Is it difficult for you to do your | Qualitative, | Proportions, frequencies, | | | |
| usual sport/leisure activity? | Ordinal | column and row totals, | | | X |
| (Variable(s): SPRACT) | | missing proportion (if any). | | | |
| | | Case summary with number | | | |
| | | and percentage of valid | X | | |
| | | cases/values, missing | | | |
| | | cases/values (if any) and total | | X | |
| ASES Pain Score [points] | Quantitative, | cases/values. | | | |
| (Variable(s): PAINSC) | ratio | Mean, median, interquartile | | | |
| | | range, maximum, minimum, | | | |
| | | standard deviation, 95% | | | |
| | | confidence interval for mean, | | | |
| | | Shapiro-Wilk Test. | ļ | | |
| | | Case summary with number | | | |
| | | and percentage of valid | | | |
| | | cases/values, missing | | | |
| AGROR C. C. C. C. | | cases/values (if any) and total | | | |
| ASES Functioning Score [points] | Quantitative, | cases/values. | X | X | |
| (Variable(s): FUNSCORE) | ratio | Mean, median, interquartile | | | |
| | | range, maximum, minimum, | | | |
| | | standard deviation, 95% | | | |
| | | confidence interval for mean, | | | |
| | | Shapiro-Wilk Test. | | | |
| | | Case summary with number | | | |
| | | and percentage of valid | | | |
| | | cases/values, missing | | | |
| The Language Line of the control of | | cases/values (if any) and total | | | |
| Total ASES Shoulder Score [points] | Quantitative, | cases/values. | X | X | |
| (Variable(s): FINSCORE) | ratio | Mean, median, interquartile | 1 | 1 | |
| | | range, maximum, minimum, | | | |
| | | standard deviation, 95% | | | |
| | | confidence interval for mean, | | | |
| | | Shapiro-Wilk Test. | | | |

Table 6.5.2: Postoperative Visit Form – ASES Shoulder Score Tables List

| Evaluation<br>Variable / Question | Level of<br>Measurement | Analysis Plan | Inclusion | | n |
|---|---|---|---|---|---|
| Postoperative Visit Form – Range of Motion | | | | FR | N/A |
| Flexion<br>(Variable(s): FLEX) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Abduction<br>(Variable(s): ABDC) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |

| Extension<br>(Variable(s): EXTN) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X |
|---|---|---|---|
| External Rotation<br>(Variable(s): EXROT) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X |
| Internal Rotation<br>(Variable(s): INTOR) | Qualitative,<br>nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X |

Table 6.5.3: Postoperative Visit Form – ROM Tables List

| Evaluation | Level of | Analysis Plan | I | nclusio | n <b>n</b> |
|---|---|---|---|---|---|
| Variable / Question | Measurement | | | | |
| Postoperative Visit Form – Rad | <u>iographic Evalua</u> | | IR | FR | N/A |
| Implant dislocation (complete dislocation) (Variable(s): QA) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Periprosthetic fracture of the humerus (Variable(s): QB) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Periprosthetic fracture of the glenoid<br>(Variable(s): QC) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Implant component dissociation<br>(humeral head from humeral stem)<br>(Variable(s): QD) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiologic signs of erosion of the glenoid (in hemiarthroplasty only) (Variable(s): QE) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Breakage of the humeral stem<br>(Variable(s): QF) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiologic signs of breakage of the glenoid component (Variable(s): QG) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiologic signs of wear of the<br>glenoid component<br>(Variable(s): QH) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiologic signs of rotator cuff tear (superior/cranial migration) (Variable(s): QI) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Heterotopic ossification<br>(Variable(s): QJ) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiolucency of the humerus<br>(Variable(s): QK) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiologic signs of gross loosening of<br>the humeral stem<br>(Variable(s): QL) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Radiolucency of the glenoid<br>(Variable(s): QM) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Gross loosening of the glenoid component (Variable(s): QN) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Non-union of lesser tuberosity<br>osteotomy<br>(Variable(s): QO) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Malunion of lesser tuberosity<br>osteotomy<br>(Variable(s): QP) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | | X | |
| Other<br>(Variable(s): QQ) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | | X | |

| Other description | Qualitative, | Listing of given description. | | X |
|---|---|---|---|---|
| (Variable(s): DESC) | Nominal | | | |
| Heterotopic ossification (modified<br>BROOKER grading)<br>(Variable(s): QS; QTG0; QTG1;<br>GR1ZN; QTG2, GR2ZN; QTG3,<br>GR3ZN; QTG4; GR4ZN; QTG5) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |
| Radiolucent lines 2 mm or greater in ≥ 3 zones (Variable(s): QU) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |
| Tilting (> 5°) or subsidence (> 5 mm)<br>of the stem<br>(Variable(s): QV) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |
| Thinning ("scalloping") of the humeral cortex (Variable(s): QW; QX) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). Listing of given description. | X | |
| Description of Radiolucency<br>(Variable(s): QY) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |
| If pegged glenoid component (Variable(s): QZ) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |
| If keeled glenoid component (Variable(s): QAA) | Qualitative,<br>Nominal | Proportions, frequencies, column and row totals, missing proportion (if any). | X | |

Table 6.5.4: Postoperative Visit Form – Radiographic Evaluation Tables List

### 6.6. ANALYSIS OF CI ENDPOINTS

| Evaluation | Level of | Analysis Plan |
|------------------------------|-------------|-----------------|
| Variable / Question | Measurement | Alialysis Flaii |
| Endpoints – Primary Endpoint | | |

Use variable Total ASES Shoulder Score 24 Months [points]:

Based on the underlying distribution of the data and the result of the normality assessment, either the parametric one-sample t-test or the non-parametric one-sample sign test will be used to compare the 24 months postoperative ASES Shoulder Score results of the ReUnion TSA group against the lower maximum acceptable difference (- $\theta$ ) of 65.40 points.

The analysis of the primary endpoint will be part of the final report.

Table 6.6.1: Endpoints – Primary Endpoint Tables List

| Evaluation<br>Variable / Question | | | | | Inclusion |
|---|---|---|---|---|---|
| Adverse Events – Time to (earlies<br>Incident | IR | FR | N/A | | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of First Device Related Adverse Event [dd.mm.yyyy] in [ days J (Variable(s): VISITDT; AEONSTDT) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. | | X | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of "most recent" Visit [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT) | | N/A (Analyzed above), used for survivorship | | X | |

| Create new variable "Grouping variable – First Device Related Adverse Event" (Variable(s): AEONSTDT) | Qualitative,<br>nominal | - censored = survivors<br>- events = first (earliest) Device<br>Related Adverse Event | X |
|---|---|---|---|
| Create new variable "Combined Time – First Device Related Adverse Event" (Variable(s): AEONSTDT) | Quantitative, ratio | - Use time between surgery and "most recent" visit for surviving subjects - Use time between surgery and first device related adverse event for subjects with device related adverse event | X |
| Use variables "Combined Time – First<br>Device Related Adverse Event"<br>and "Grouping variable – First Device<br>Related Adverse Event" | Qualitative,<br>nominal<br>Quantitative,<br>ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Kaplan-Meier survival analysis: subject ID, time, status, cumulative proportion, Kaplan-Meier estimate, standard error of KM estimate, number of cumulative events, number of remaining cases, mean for survival time with 95% confidence interval, survival graph, hazard graph. | X |

Table 6.6.2: Endpoints – Secondary Endpoint Time to (earliest) Device Related Adverse Event / Incident Tables List

### 6.7. ADDITIONAL ANALYSIS

### 6.7.1. ASES Comparison

The comparison of the ASES Shoulder Score must compare all Total ASES Shoulder Scores of all follow-up visits against each other  $(m \times n)$  in accordance to table 6.7.1.1 and the analysis tables listed in this chapter. This analysis is part of the final report only.

| | ASES Shoulder Score – Follow-up Visits to be compared | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Follow-up Visits (n) | | | | | | | | | | | |
| Comparison | | Preop | 6 Weeks | 6 Months | 12 Months | 24 Months | 36 Months | 48 Months | 60 Months | 72 Months | 84 Months | 96 Months | 108 Months | 120 Months |
| | Preop | | | | | | | | | | | | | |
| | 6 Weeks | X | | | | | | | | | | | | |
| | 6 Months | X | X | | | | | | | | | | | |
| m) | 12 Months | X | X | X | | | | | | | | | | |
| B ( | 24 Months | X | X | X | X | | | | | | | | | |
| sits | 36 Months | X | X | X | X | X | | | | | | | | |
| Follow-up Visits B (m) | 48 Months | X | X | X | X | X | X | | | | | | | |
| dn-/ | 60 Months | X | X | X | X | X | X | X | | | | | | |
| llow | 72 Months | X | X | X | X | X | X | X | X | | | | | |
| Fo | 84 Months | X | X | X | X | X | X | X | X | X | | | | |
| | 96 Months | X | X | X | X | X | X | X | X | X | X | | | |
| | 108 Months | X | X | X | X | X | X | X | X | X | X | X | | |
| | 120 Months | X | X | X | X | X | X | X | X | X | X | X | X | |
| *All | combinations marked | with | an "x" | must | be perf | formed | | | | | | | | |

Table 6.7.1.1: All Assessments – ASES Shoulder Score – Follow-up Visits to be compared

| Evaluation | Level of | Analysis Dlan |
|---|---|---|
| Variable / Question | Measurement | Analysis Plan |
| All Assessments – ASES Shoulder Score Comparison | | |
| | Use "ASES Total Score m [points]" and "ASES Total Score n [points]": | |
| Based on the underlying distribution | of the data in both gro | oups and the result of the normality assessment, either |
| the parametric paired samples t-test | or the non-parametric | Wilcoxon test will be used to compare |
| "ASES Total Score m [points]" and | "ASES Total Score n | [points]" to evaluate the ASES Shoulder Score |
| change by subject (improvement or o | decrease). | |
| The complete available SPSS tables | content related to eithe | er the paired samples t-test or the Wilcoxon test will |
| be included in the final report. | | |
| (Variable(s): FINSCORE) | | |

Table 6.7.1.2: All Assessments – ASES Shoulder Score Comparison Tables List

### 6.7.2. Mortality

For analysis of the time to death or mortality, the Kaplan-Meier method will be used. The times between surgery and the most recent or last available assessment per subject will be used together with the times between surgery and the date of death. This analysis is part of the final report.

| Evaluation<br>Variable / Question | Level of<br>Measurement | Recode and Analysis Plan |
|---|---|---|
| All Assessments – Mortality | | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of Death [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT; DOSEDD) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean. Shapiro-Wilk Test. |

| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of "most recent" Visit [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT) | Quantitative, ratio | N/A (Analyzed above), used for survivorship |
|---|---|---|
| Create new variable "Grouping variable -<br>Mortality"<br>(Variable(s): PRIMRSN) | Qualitative,<br>nominal | - censored = survivors<br>- events = death |
| Create new variable "Combined Time -<br>Mortality"<br>(Variable(s): VISITDT; DOSEDD) | Quantitative, ratio | Use time between surgery and most recent visit for surviving subjects Use time between surgery and death for deceased subject |
| Use variables "Combined Time -<br>Mortality" and "Grouping variable -<br>Mortality" | Qualitative,<br>nominal<br>Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Kaplan-Meier survival analysis: subject ID, time, status, cumulative proportion, Kaplan-Meier estimate, standard error of KM estimate, number of cumulative events, number of remaining cases, mean for survival time with 95% confidence interval, survival graph, hazard graph. |

Table 6.7.2.1: All Assessments – Mortality Tables List

### 6.7.3. Reoperation Surgery

For analysis of the time to the reoperation surgery, the Kaplan-Meier method will be used. The times between surgery and the most recent or last available assessment per subject will be used together with the times between surgery and the date of reoperation (earliest reoperation in case that one subject experienced more than one reoperation). This analysis is part of the final report.

| Evaluation | Level of | |
|---|---|---|
| Variable / Question | Measurement | Recode and Analysis Plan |
| Adverse Events / Reoperation S | urgery | |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of First Reoperation [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT) | Quantitative, ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |
| Creation of variable Difference between Date of Surgery [dd.mm.yyyy] and Date of "most recent" Visit [dd.mm.yyyy] in [ days ] (Variable(s): VISITDT) | Quantitative, ratio | N/A (Analyzed above), used for survivorship |
| Create new variable "Grouping variable - First Reoperation" (Variable(s): VISITDT) | Qualitative,<br>nominal | - censored = survivors<br>- events = first (earliest) Reoperation |
| Create new variable "Combined Time – First Reoperation" (Variable(s): VISITDT) | Quantitative, ratio | <ul> <li>Use time between surgery and most recent visit for surviving subjects</li> <li>Use time between surgery and first reoperation for subjects with reoperation(s)</li> </ul> |
| Use variables "Combined Time – First<br>Reoperation" and "Grouping variable –<br>First Reoperation" | Qualitative,<br>nominal<br>Quantitative,<br>ratio | Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Kaplan-Meier survival analysis: subject ID, time, status, cumulative proportion, Kaplan-Meier estimate, standard error of KM estimate, number of cumulative events, number of remaining cases, mean for survival time with 95% confidence interval, survival graph, hazard graph. |

Table 6.7.3.1: All Assessments – Reoperation Surgery Tables List

### 6.7.4. ASES Shoulder Score – Within subject changes by visit

The within subject score changes of the ASES Shoulder Score from visit to visit will be analyzed to help identifying the changes on the subject level. This analysis is part of the final report.

The within subject changes by visit of the ASES Shoulder Score must compare all follow-up visits against each other  $(m \times n)$  in accordance to table 6.7.4.1 and the analysis tables in this chapter.

| ASES Shoulder Score – Follow-up Visits to be compared | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Follow-up Visits (n) | | | | | | | | | | | | | |
| ( | Comparison | Preop 6 Weeks 6 Months 12 Months 36 Months 48 Months 72 Months 84 Months 96 Months | | | | | | 108 Months | 120 Months | | | | |
| | Preop | | | | | | | | | | | | |
| | 6 Weeks | X | | | | | | | | | | | |
| | 6 Months | X | X | | | | | | | | | | |
| m) | 12 Months | X | X | X | | | | | | | | | |
| B ( | 24 Months | X | X | X | X | | | | | | | | |
| sits | 36 Months | X | X | X | X | X | | | | | | | |
| Vi | 48 Months | X | X | X | X | X | X | | | | | | |
| n | 60 Months | X | X | X | X | X | X | X | | | | | |
| Follow-up Visits B (m) | 72 Months | X | X | X | X | X | X | X | X | | | | |
| Fol | 84 Months | X | X | X | X | X | X | X | X | X | | | |
| | 96 Months | X | X | X | X | X | X | X | X | X | X | | |
| | 108 Months | X | X | X | X | X | X | X | X | X | X | X | |
| | 120 Months | X | X | Х | X | X | X | X | X | X | X | X | X |
| *All | combinations marked | with | an "x" | must | be per | formed | | | | | | | |

Table 6.7.4.1: All Assessments – ASES Shoulder Score – Follow-up Visits to be compared

| | Level of<br>Measurement | Coding and Analysis Plan |
|---|---|---|
| All Assessments - ASES Shoulder Score Within Subject Changes | | |
| Creation of variable "ASES Total Score change between m and n [points]" Difference between "ASES Total Score m [points]" with "ASES Total Score n [points]" (Variable(s): FINSCORE) | Quantitative, interval | Calculate difference (could be negative or positive). Case summary with number and percentage of valid cases/values, missing cases/values (if any) and total cases/values. Mean, median, interquartile range, maximum, minimum, standard deviation, 95% confidence interval for mean, Shapiro-Wilk Test. |

Table 6.7.4.2: All Assessments – ASES Shoulder Score Within Subject Changes

### 7. Table Templates (Tables, Figures, Listings - TFL)

Tables must consist of at least a headline, the variable/analysis-object label and column headers. Furthermore, the table headline must contain the "Analysis Section" (e.g. Demographics, Operative) the variable label (e.g. Gender, Age) as well as the table type (Frequencies, Listing). If the table is referring to a subgroup, a notification must be entered in the headline as well. Figures (if any) must be clearly labeled and numbered by a figure number and title in addition to the axis and category labeling created by software packages (e.g. IBM SPSS).

#### 7.1. FREQUENCIES

All answered response options must be listed with the appropriate label, other response options do not have to be displayed necessarily. In the event of missing answers, the frequencies must be included in an extra row as well ("Missing"). All given answers must be added up in an extra row ("Total"). In addition to the number of frequencies, percentages must be displayed in a separate column.

"Analysis Section" - "Variable Label" - Frequencies

| Characteristic | | n | % |
|------------------|--------------|-------|-------|
| | "Response A" | "xxx" | "xxx" |
| "I/: | "Response B" | "xxx" | "xxx" |
| "Variable Label" | Missing | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" |

Table 7.1.1: Frequencies Table Template

If multiple subgroups/clusters (e.g. Sites, Visits) should be displayed in one table, an extra column ("Group X") and/or extra rows ("Group Y") must be added. Same applies to (sub-) questions, which can be merged in one table. It is recommended to add an extra "Total" column and row, for adding up the subgroups, if possible, from a statistical point of view. In addition, subgroups must be named in the headline as well ("by Group X and by Group Y").

"Analysis Section" – "Variable Label" – Frequencies – by "Group X" and "Group Y"

| Chamatanistic | | "Grou | p X1" | "Grou | ıp X2" | Total | |
|---|---|---|---|---|---|---|---|
| Characteristi | Characteristic | | % | n | % | n | % |
| | "Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Curry VI" | "Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Group Y1" | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | "Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Group V2 | "Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| "Group Y2 | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | "Total Response A" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| Total | "Total Response B" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| Total | Missing | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |
| | Total | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" | "xxx" |

Table 7.1.2: Grouped Frequencies Table Template

#### 7.2. DESCRIPTIVE STATISTICS

Descriptive Statistic tables must contain the items listed in Table 7.2.1. Furthermore, the associated unit must be displayed. If the values are referring to a subgroup (n) and not to the overall population (N), a notification must be entered in the headline ("n = xxx").

### "Analysis Section" – "Variable Label" – Descriptive Statistics (n = "xxx")

| Characteristic | | ["unit"] |
|------------------|--------|----------|
| "Variable Label" | Mean | "xxx" |
| | Median | "xxx" |
| | SD | "xxx" |
| | IQR | "xxx" |
| | Range | "xxx" |
| | Max | "xxx" |
| | Min | "xxx" |

Table 7.2.1: Descriptive Statistics Table Template

### 7.3. LISTINGS

Listing tables must contain one unique identifier (e.g. Subject ID). Furthermore, an additional column must be added, if the specification/description is not referring to one single variable or response option("Response Option"), which is already named in the headline. If multiple specifications/descriptions exist for one variable/response (e.g. Drug1, Drug2, Drug3...), further columns must be added ("Specification/Description A", "Specification/Description B"). Subgroups can be implemented as described in chapter 7.1.

### "Analysis Section" - "Variable Label" - Listing

| "Unique | Description | |
|-------------|-------------------|-------------------------------|
| Identifier" | "Response Option" | "Specification/Description A" |
| "xxx" | "xxx" | "xxx" |
| "xxx" | "xxx" | "xxx" |
| "xxx" | "xxx" | "xxx" |

Table 7.3.1: Listing Table Template

### 8. References

- a. ISO 14155 Clinical Investigation of Medical Devices for Human Subjects
- b. ICH-E6 Harmonized Tripartite Guidelines for Good Clinical Practice
- c. ICH-E9 Statistical Principles for Clinical Trials
- d. Declaration of Helsinki
- e. Gamble C et. al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. AMA. 2017;318(23):2337-2343. doi:10.1001/jama.2017.18556
- f. DQP 20-001 Clinical Investigation
- g. DQI 20-001 Clinical Investigation Clinical Investigation Plan
- h. DQI 20-004 Clinical Investigation Master CRF, eCRF and Database Development
- i. DQI 20-009 Clinical Investigation Reports

# 20210528\_ReUnion TSA\_SAP

Final Audit Report 2021-05-28

Created: 2021-05-28

By: Sascha Lorenzen (sascha.lorenzen@stryker.com)

Status: Signed

Transaction ID: CBJCHBCAABAAdMdB-jSdyk8ccXhiXIY6GCjnoGnlruGD

# "20210528\_ReUnion TSA\_SAP" History

- Document created by Sascha Lorenzen (sascha.lorenzen@stryker.com) 2021-05-28 11:47:37 AM GMT- IP address: 46.114.169.5
- Document emailed to Sascha Lorenzen (sascha.lorenzen@stryker.com) for signature 2021-05-28 11:49:31 AM GMT
- Document emailed to Rebecca Gibson (rebecca.gibson@stryker.com) for signature 2021-05-28 11:49:31 AM GMT
- Document emailed to Claudia Beimel (claudia.beimel@stryker.com) for signature 2021-05-28 11:49:31 AM GMT
- Document emailed to Susanne Höfer (susanne.hoefer@stryker.com) for signature 2021-05-28 11:49:31 AM GMT
- Sascha Lorenzen (sascha.lorenzen@stryker.com) verified identity with Adobe Sign authentication 2021-05-28 11:50:34 AM GMT
- Document e-signed by Sascha Lorenzen (sascha.lorenzen@stryker.com)

  Signature Date: 2021-05-28 11:50:34 AM GMT Time Source: server- IP address: 46.114.169.5
- Email viewed by Rebecca Gibson (rebecca.gibson@stryker.com) 2021-05-28 12:29:13 PM GMT- IP address: 52.154.71.15
- Rebecca Gibson (rebecca.gibson@stryker.com) verified identity with Adobe Sign authentication 2021-05-28 - 12:31:23 PM GMT
- Document e-signed by Rebecca Gibson (rebecca.gibson@stryker.com)
  Signature Date: 2021-05-28 12:31:23 PM GMT Time Source: server- IP address: 52.154.71.15
- Claudia Beimel (claudia.beimel@stryker.com) verified identity with Adobe Sign authentication 2021-05-28 - 12:37:09 PM GMT



Document e-signed by Claudia Beimel (claudia.beimel@stryker.com)

Signature Date: 2021-05-28 - 12:37:09 PM GMT - Time Source: server- IP address: 159.100.98.130

Email viewed by Susanne Höfer (susanne.hoefer@stryker.com) 2021-05-28 - 1:28:23 PM GMT- IP address: 91.58.232.30

- Susanne Höfer (susanne.hoefer@stryker.com) verified identity with Adobe Sign authentication 2021-05-28 1:30:01 PM GMT
- Document e-signed by Susanne Höfer (susanne.hoefer@stryker.com)

  Signature Date: 2021-05-28 1:30:01 PM GMT Time Source: server- IP address: 91.58.232.30
- Agreement completed. 2021-05-28 - 1:30:01 PM GMT